CLINICAL TRIAL: NCT05771012
Title: Topical Cyclosporin A 0.05% Eye Drops for Management of Symptomatic Acquired Punctal Stenosis. A Prospective, Controlled Clinical Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Nancy Lotfy, MD, Dr, Farwaniya Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1482
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Management of Punctal Stenosis
Keywords: cyclosporin,; punctal stenosis,; Restasis,; mini-Monoka.
MeSH Terms: interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group A (Experimental): patients receive only medical treatment in the form of topical 0.05% cyclosporin (Restasis®, Allergan Inc) twice daily for 6 months.
  Interventions: Drug: 0.05% cyclosporin (Restasis®, Allergan Inc)
- group B (Active Comparator): patients receive mini-Monoka stent insertion in the lower canaliculus for 6 months.
  Interventions: Device: mini-monoka stent

INTERVENTIONS:
Drug: 0.05% cyclosporin (Restasis®, Allergan Inc) — study the efficacy of topical 0.05% cyclosporin eye drops (Restasis®, Allergan Inc) in management of grade 1 and 2 acquired punctal stenosis (group A)
  Arms: group A
Device: mini-monoka stent — insertion of mini-monoka stent in the lower punctum in management of grade 1 and 2 acqquired punctal stenosis (group B)
  Arms: group B

SUMMARY:
A prospective, controlled, interventional clinical study, includes all patients (16 years) with symptomatic epiphora and diagnosed with grade 1 or grade 2 acquired punctal stenosis. All patients undergo punctal dilatation, canalicular probing and nasolacrimal duct irrigation. Afterwards, patients are divided into two groups: Group A: patients receive only medical treatment in the form of topical 0.05% cyclosporin (Restasis®, Allergan Inc) twice daily for 6 months. Group B: patients receive mini-Monoka stent insertion in the lower canaliculus for 6 months. Outcome measures are changes in Munk scoring, grading of the punctum, functional and anatomical success. Functional success is defined as Munk score 0 to 1. Anatomical success is defined as grade 3 punctum.

ELIGIBILITY:
Inclusion Criteria:

* The study includes all patients (more than 16 years) with symptomatic epiphora and diagnosed with grade 1 or grade 2 acquired punctal stenosis

Exclusion Criteria:

* Patients presented with congenital epiphora, previous eyelid surgeries, neoplastic or traumatic causes of punctual or canalicular obstruction, or any other causes of lacrimal passage obstruction such as canalicular, common canalicular or nasolacrimal duct obstruction NLDO are excluded from this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
functional success | 6 months
  change in munk score
anatomical success | 6 months
  grading of the punctum by measuring its size in millimeters on slit lamp

CONTACTS AND LOCATIONS:
Overall Officials: Mona Nassief, Principal Investigator — Farwaniya Hospital
Locations (1):
- Farwanyia Hospital, Al Farwānīyah, Farwanyia, Kuwait